CLINICAL TRIAL: NCT02704078
Title: Prospective Randomized Comparison of Trans-tracheal (EBUS-TBNA) Versus Trans-esophageal (EUS-B-FNA) Route as the Primary Approach for Fine Needle Aspiration of Mediastinal Lesions Using the Convex Probe Endobronchial Ultrasound (EBUS) Scope
Brief Title: EBUS-TBNA vs EUS-B-FNA for Needle Aspiration of Mediastinal Lesions
Acronym: TEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Karan Madan, Dr. Karan Madan, MD, DM Assistant Professor, Pulmonary MedicIne and Sleep Disorders, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IEC/NP-419/09.10.2015
Record Dates: First submitted 2016-02-25; First posted 2016-03-09 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Mediastinum

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EBUS-TBNA (Active Comparator): Mediastinal lymph node aspiration shall be performed transtracheally.
  Interventions: Device: EBUS-TBNA
- EUS-B-FNA (Experimental): Mediastinal lymph node aspiration shall be performed transesophageally
  Interventions: Device: EUS-B-FNA

INTERVENTIONS:
Device: EBUS-TBNA — EBUS-TBNA - Patients in the Active comparator arm shall undergo mediastinal lymph node aspiration transtracheally using the EBUS scope
  Arms: EBUS-TBNA
Device: EUS-B-FNA — EUS-B-FNA - Patients in the experimental arm EUS-B-FNA shall undergo mediastinal lymph node aspiration transesophageally using the EBUS scope
  Arms: EUS-B-FNA

SUMMARY:
Endobronchial Ultrasound Guided Transbronchial Needle aspiration (EBUS-TBNA) is a firmly established modality for diagnostic evaluation of mediastinal lesions. The procedure is routinely performed at the Department of Pulmonary Medicine and Sleep Disorders, AIIMS, New Delhi since 2012. Transesophageal approach for fine needle aspiration of mediastinal lesions using the Endobronchial Ultrasound (EBUS) scope [also described as Transesophageal Bronchoscopic Ultrasound Guided Fine Needle aspiration (EUS-B-FNA)] (also routinely performed in the department) and has been described as a safe and efficacious modality. EUS-B-FNA is usually employed when EBUS-TBNA is not feasible or excessive cough or secretions necessitate switch to esophageal route. We hypothesize that EUS-B-FNA as the primary approach has similar diagnostic performance as EBUS-TBNA and is associated with greater patient and operator rated procedure comfort and lesser requirement of anaesthesia medications for evaluation of patients with mediastinal lesions easily accessible with either of the two approaches.

We propose to undertake a prospective randomized comparison of Transesophageal (EUS-B-FNA) versus Transtracheal (EBUS-TBNA) approach for fine needle aspiration using the same EBUS scope in patients referred for endo-sonographic evaluation of mediastinal lesions. A total of 100 serial patients (with Subcarinal and/or Lower Left paratracheal located mediastinal lymphadenopathy at least >1cm in Short axis diameter) shall be included. After consent and preliminary investigations, patients shall be randomized equally into the two approaches. Procedure will be performed under local anaesthesia (topical lignocaine) and i.v. sedation (midazolam and fentanyl) in the bronchoscopy laboratory. The primary objective will be comparison of proportion of diagnostic and adequate aspirates in the two groups. Secondary objectives will include operator rated cough (VAS), Operator rated overall procedure satisfaction (VAS), dose of midazolam and fentanyl administered, lignocaine dose and total procedure duration.The primary data analysis shall be for the performance characteristics of the primary approach. All the aspirates shall be analysed by the same pathologist for final interpretation.

DETAILED DESCRIPTION:
Objectives

Primary objective:

Comparison of Proportion of Adequate and Diagnostic Aspirates in the EUS-B-FNA versus EBUS-TBNA arms as the primary approach for mediastinal fine needle aspiration during Convex probe EBUS.

Secondary objectives

1. Topical Anaesthetic requirement between the two groups
2. Intravenous Sedative / analgesic requirement between the two groups
3. Operator rated overall procedure satisfaction (VAS)
4. Operator rated cough (VAS)
5. Overall duration of procedure Methods Study Design: Prospective randomised study. Sample Size: Number of Patients: 100 (50 -EBUS-TBNA arm, 50- EUS-B-FNA arm)

Inclusion criteria:

* Age 18 years and Older
* Patients with predominant Subcarinal or Lower Left paratracheal located mediastinal lymphadenopathy/mediastinal lesions at least >1cm in Short axis diameter.
* Patients who give consent.

Exclusion criteria:

* Refusal of consent for the procedure
* Any contraindications to Bronchoscopy or Endobronchial Ultrasound procedures
* Pregnancy Controls: None For all patients, a targeted history will be obtained to screen for diabetes mellitus, systemic hypertension, bleeding disorders, cardiac disease, previous anaesthetic complications and any medication history including antiplatelet therapy. Baseline investigations like complete hemogram and prothrombin time will be done, and imaging prior to the procedure will include a chest radiograph and computed tomography (CT) scan of the chest (plain and contrast enhanced).

The patients will then be randomised to 2 groups of 50 patients each. 50 patients in one group will undergo Transtracheal (EBUS-TBNA) approach, whereas in the other group, 50 patients will undergo Transesophageal (EUS-B-FNA) route as the primary approach using the EBUS scope. Procedures will be performed under moderate sedation. Procedures will be performed in the Bronchoscopy Lab.

The size and characteristics of the mediastinal lymph nodes as visualised during EBUS/EUS will be recorded. The concerned mediastinal lymph nodes will be sampled by EBUS-TBNA/EUS-FNA under direct ultrasonic visualisation. The aspirates will be expressed on to slides and will be placed into alcohol cytology bottles. The slides will then be dispatched to the Cytopathology Lab for appropriate stains and further analysis. Lymph node core if obtained will be sent in formalin for Histopathological analysis. Post procedure, the patients will remain in observation for a few hours and will be discharged on the same day. A patient proforma will be completed for each patient separately. The size and stations of the sampled nodes will be recorded. The total duration of procedure, the nature and total dose of anaesthesia or sedation will also be recorded. A Visual-analogue scale (VAS) will be used to assess operator rated procedure related cough and overall operator rated procedure satisfaction.

Statistical Analysis - Descriptive statistics such as mean, median, standard deviation and range will be calculated for all continuous variables. Frequency distributions will be calculated for all qualitative data. Frequency data across categorical variables will be compared using chi-square and fisher's exact test. Among patients with adequate sample on EBUS-TBNA/EUS-B-FNA, sensitivity, specificity, accuracy, and positive and negative predictive values will be calculated using standard formulas. P-value of P<0.05 is considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and Older
* Predominant Subcarinal or Lower Left paratracheal located mediastinal lymphadenopathy/mediastinal lesions at least >1cm in Short axis diameter.
* Patients who give consent

Exclusion Criteria:

* Refusal of consent for the procedure
* Any contraindications to Bronchoscopy / Endobronchial Ultrasound
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Diagnostic Sensitivity of EUS-B-FNA versus EBUS-TBNA | At study completion at approximately 18 months
  The diagnostic yield of EBUS-TBNA shall be compared with EUS-B-FNA ie comparison of the proportion of diagnostic aspirates between the EBUS-TBNA and the EUS-B-FNA groups

SECONDARY OUTCOMES:
Topical Anaesthetic requirement between the two groups | Comparing the mean doses of lignocaime administered in mg between the study participants in two groups at study completion at approximately 18 months
  Comparison of total lignocaine dose
Intravenous Sedative / analgesic requirement between the two groups | Compating the mean doses of sedative administered in mg between the study participants in two groups at study completion at approximately 18 months
  Comparison of midazolam/fentanyl dose
Operator rated overall procedure satisfaction (VAS) | At study completion at approximately 18 months
  Comparison of VAS scores
Operator rated cough between the two procedures (VAS) | At study completion at approximately 18 months
  Comparison of VAS scores
Overall duration of procedure | Intraoperative
  Comparison of time taken

CONTACTS AND LOCATIONS:
Overall Officials: Randeep Guleria, Study Chair — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided